CLINICAL TRIAL: NCT05651867
Title: Prospective Clinical Investigation on the Evaluation of Performance and Safety of the EPIONE Assisted CT-guided Percutaneous Procedures in the Lungs
Brief Title: EPIONE Guided Lung Evaluation
Acronym: EGLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quantum Surgical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QS-IS-G-H-2201
Record Dates: First submitted 2022-11-28; First posted 2022-12-15 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
Keywords: percutaneous; CT-guided; Ablation; Biopsy; Abcess Drainage; Fiducial placement; Lung; Robotics
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interventional arm (Experimental): Patients treated by percutaneous CT-guided procedures in the lung with the EPIONE® device
  Interventions: Device: EPIONE device

INTERVENTIONS:
Device: EPIONE device — The EPIONE device is a user controlled, stereotactic accessory intended to assist in the planning and manual advancement of one or more instruments, as well as in verification of instrument position during Computed Tomography (CT) guided percutaneous procedures.

SUMMARY:
Interventional clinical study to obtain performance and safety data of the EPIONE® device when used for percutaneous procedures in the lung.

DETAILED DESCRIPTION:
The objectives are:

* to evaluate the technical success of the device
* to evaluate performance parameters (accuracy measures, adjustements, post-intervention ablation success, local tumor recurrence)
* to evaluate the safety of the device

  25 subjectsare planned and will undergo an intervention, during which the clinician will use the EPIONE device

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥18 years old,
* Patient for whom a percutaneous CT-guided intervention in lung has been prescribed and agreed by a multidisciplinary team of radiologists, surgeons and clinicians,
* Patient with a signed informed consent form.
* Patient covered by a social security system.

Exclusion Criteria:

* Patient unable to undergo general anesthesia,
* Pregnant or nursing female, confirmed before the intervention
* Patient already participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2024-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baptiste BONNET, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy Institut, Villejuif, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 25 patients included from 2022-11-30 to 2023-08-25 at the IGR (Villejuif/France).
Period: Overall Study
Arm/Group | Interventional Arm
Started | 25
Completed | 19
Not Completed | 6

BASELINE CHARACTERISTICS:
Population: number of lesions treated with the Epione device
Units Other Than Participants: lesions
Arm/Group | Interventional Arm
Number analyzed (Participants) | 25
Number analyzed (lesions) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 25.2 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Device
Description: Number of lesion target reached ; the lesion target is considered reached when the needle is positioned accurately enough as compared to the planning to allow the planned procedure to be performed.
Time Frame: an average of 7 months
Population: All screened patients who have confirmed their signed informed consent and are planned to be treated using the EPIONE® device.
Measure: Count of Units; unit: Number of targets reached
Units Other Than Participants: Number of targets reached
Arm/Group | Interventional Arm
Number analyzed (Participants) | 25
Number analyzed (Number of targets reached) | 27
Number of targets reached | 26

2. Secondary Outcome: Needle Placement Accuracy
Description: accuracy of the needle placement: deviation between the planned and actual needle position once inserted.
Time Frame: an average of 7 months
Population: all patients whose procedure was feasible
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: needles
Arm/Group | Interventional Arm
Number analyzed (Participants) | 24
Number analyzed (needles) | 30
mm | 1.2 (2.1)

3. Secondary Outcome: Number of Needle Adjustments
Description: Detail of the number/nature of adjustments performed after the initial insertion of the needle.
Time Frame: an average of 7 months
Population: all patients whose procedure was feasible
Measure: Mean (Standard Deviation); unit: number of adjustments per needle
Units Other Than Participants: needle
Arm/Group | Interventional Arm
Number analyzed (Participants) | 24
Number analyzed (needle) | 30
number of adjustments per needle | 0.8 (0.5)

4. Secondary Outcome: Post-intervention Ablation Success
Description: If the ablation zone is at least the lesion size + 5mm, the ablation is considered successfull. The measure counted is the number of success
Time Frame: an average of 1 year
Population: all patients whose procedure was feasible
Measure: Count of Units; unit: lesions
Units Other Than Participants: lesions
Arm/Group | Interventional Arm
Number analyzed (Participants) | 24
Number analyzed (lesions) | 26
lesions | 20

5. Secondary Outcome: Long-term Efficacy of Ablation
Description: If a tumor progresses locally 12 months after the initial treatment, the long-term efficacy of the ablation is considered failed.
  We count here the patient treated for which the lesion ablated did not show recurrence after 12 months.
Time Frame: through study completion, an average of 1 year
Population: all patients whose procedure was feasible and were still in the study after 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 19
Participants | 18

6. Secondary Outcome: Adverse Event
Description: number of patients experiencing a serious adverse event
Time Frame: through study completion, an average of 21 months
Population: all patients included in the study
Measure: Number; unit: participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 25
participants | 5

7. Secondary Outcome: Grade of Needle Adjustment
Description: Description of the grade of needle adjustement : minor meaning depth needle adjustment only, medium meaning at lateral needle adjustement (+ or - depth adjustement) or major (meaning complete removal of the needle from the atient body)
Time Frame: an average of 7 months
Population: all patients who started the procedure with EPIONE
Measure: Count of Units; unit: needle
Units Other Than Participants: needle
Arm/Group | Interventional Arm
Number analyzed (Participants) | 25
Number analyzed (needle) | 31
needle
  minor adjutsments | 7
  medium adjustements | 17
  major adjustements | 1
  no adjustement | 6

ADVERSE EVENTS:
Time Frame: through study completion, an average of 21 months
Arm/Group | Interventional Arm
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 8/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm (N=25)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 4 (4)
ABCESS (Infections and infestations) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumapathy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interventional Arm (N=25)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Haemorrhage (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-05-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT05651867/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/67/NCT05651867/SAP_001.pdf